CLINICAL TRIAL: NCT00403650
Title: Inhaled Iloprost for Sarcoidosis Associated Pulmonary Hypertension
Brief Title: Inhaled Iloprost for Sarcoidosis-associated Pulmonary Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Robert P Baughman, Professor of Medicine, University of Cincinnati
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sarcoid 6
Record Dates: First submitted 2006-11-24; First posted 2006-11-27 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-04

CONDITIONS: Sarcoidosis; Pulmonary Arterial Hypertension
Keywords: Sarcoidosis; Dyspnea; Interstitial lung disease
MeSH Terms: conditions — Sarcoidosis; Pulmonary Arterial Hypertension; Dyspnea; Lung Diseases, Interstitial | interventions — Iloprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Iloprost

INTERVENTIONS:
Drug: Iloprost — Iloprost 2.5-5 mg inhaled via nebulizer up to 6 times a day
  Other Names: Ventavis

SUMMARY:
This trial will study the treatment of sarcoidosis-associated pulmonary arterial hypertension with inhaled iloprost, a drug approved for primary pulmonary arterial hypertension.

DETAILED DESCRIPTION:
Pulmonary hypertension has been described in sarcoidosis. It can be a significant problem, not responsive to treatment with anti-inflammatory drugs for the sarcoidosis (1;2). Inhaled iloprost has been approved for treatment of pulmonary hypertension (3). We propose to study the effectiveness of inhaled iloprost for sarcoidosis associated pulmonary hypertension (SAPAH). This is an open label trial, with patients receiving 16 weeks of therapy. Clinical and hemodynamic outcome of therapy will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known sarcoidosis 17
* Age 18 or greater
* Patients with documented pulmonary hypertension with a PA mean > 25 mm as measured by cardiac catheterization within six months of entry into the study
* Patients with dyspnea
* Six minute walk distance of between 100 to 500 meters
* Patients on stable immunotherapy for their sarcoidosis, including prednisone, methotrexate, azathioprine, hydroxychloroquine, cyclophosphamide, thalidomide, and/or infliximab
* Patients able to provide written consent

Exclusion Criteria:

* Patients on pulmonary vasodilator drugs (flolan, remodulin, bosentan, sildenafil) in the prior 28 days (patients on stable dose of calcium channel blocker for more than 1 month prior to right heart catheterization can be continued on the calcium channel blocker)
* Patients with severe airway obstruction as defined by FEV1/FVC of less than 35%
* Patients with World Health Organization (WHO) class IV status
* Patients who are pregnant or breast feeding
* Patients with significant left ventricular dysfunction with a left ventricular ejection fraction of less than 35%
* Significant liver dysfunction not due to sarcoidosis
* Patients with severe other organ disease felt by investigators to impact survival during the course of the study
* Patients unable to perform the 6 inhalation treatments required for therapy
* Patients with < 90 mm Hg Systolic systemic blood pressure will be excluded

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-11; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Change in six minute walk distance | 24 weeks

SECONDARY OUTCOMES:
Quality of life | 24 weeks
Respiratory function | 24 weeks
Toxicity | 24 weeks
Pulmonary artery hemodynamics | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert P. Baughman, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Baughman RP, Judson MA, Lower EE, Highland K, Kwon S, Craft N, Engel PJ. Inhaled iloprost for sarcoidosis associated pulmonary hypertension. Sarcoidosis Vasc Diffuse Lung Dis. 2009 Jul;26(2):110-20. PMID 20560291